CLINICAL TRIAL: NCT05507424
Title: Prone Positioning During Delayed Cord Clamping: A Randomized Control Pilot Study to Identify Optimal Neonatal Positioning During Delayed Cord Clamping
Brief Title: Prone Positioning During Delayed Cord Clamping
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: West Penn Allegheny Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00307467
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Delayed Cord Clamping
Keywords: Umbilical Cord Clamping; Preterm Birth; Delayed Cord Clamping (DCC)
MeSH Terms: conditions — Premature Birth | interventions — Prone Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prone Positioning During Delayed Cord Clamping (Active Comparator): Newborns delivered between 25w+0d and 29w+6d gestation who have been randomized in 1:1 fashion to prone positioning during routine delayed cord clamping.
  Interventions: Procedure: Prone Positioning
- Supine Positioning During Delayed Cord Clamping (Active Comparator): Newborns delivered between 25w+0d and 29w+6d gestation who have been randomized in 1:1 fashion to supine positioning during routine delayed cord clamping.
  Interventions: Procedure: Supine Positioning

INTERVENTIONS:
Procedure: Prone Positioning — Newborn will be prone position for 30-60 seconds during delayed umbilical cord clamping
  Arms: Prone Positioning During Delayed Cord Clamping
Procedure: Supine Positioning — Newborn will be supine position for 30-60 seconds during delayed umbilical cord clamping
  Arms: Supine Positioning During Delayed Cord Clamping

SUMMARY:
Delayed cord clamping is a routine technique used in the delivery room. The baby remains attached to the umbilical cord and placenta for 30-60 seconds after birth to allow for maximal transfer of oxygen and blood to the newborn. This study seeks to determine the best position (on the back versus on the belly) for the newborn during the 30-60 seconds of delayed cord clamping.

DETAILED DESCRIPTION:
This study is being done to see if placing babies on the stomach or the back during delayed cord clamping after birth will improve the outcomes of preterm babies. Studies have shown that in some instances, positioning on the belly may help newborns clear their respiratory secretions. Research has shown that preterm babies can have improved breathing and require less support when placed on the stomach (prone position) rather than the back (supine position). Currently there are no guidelines for the best position for neonates to be in while receiving delayed cord clamping. The investigators are hoping to complete a research study to determine if placing preterm babies on their stomachs during the time of delayed cord clamping will improve the breathing of preterm babies and reduce the need for additional oxygen support with a breathing tube (endotracheal intubation). Depending on the outcomes of the study, the investigators are hoping to determine which position results in better outcomes for babies in both the delivery room and in the neonatal intensive care unit. If the investigators are able to determine the optimal position in this study, the investigators hope to improve the outcomes for future babies that are born preterm by placing the baby in the optimal position during delayed cord clamping.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patient admitted for diagnosis that could result in a preterm delivery
* Anticipated gestational age of delivery could be between 25w+0d - 29w+6d
* Fetus without major anomalies or known genetic condition that could impact respiratory status or need for intubation at birth
* Singleton or twin gestation
* Neonate eligible for delayed cord clamping based on institutional protocol
* Patient is able to understand study procedures and is willing and able to consent

Exclusion Criteria:

* Triplet or higher order gestation
* Maternal or fetal/neonatal contraindication to delayed cord clamping
* Major fetal anomaly that would be expected to impact delivery room intubation rates such as:

  * Major congenital cardiac defect (not isolated atrial septal defect/ventricular septal defect)
  * Significant fetal arrhythmia at the time of delivery
  * Fetal tumor
  * Renal anhydramnios (not isolated urinary tract dilation with normal fluid)
  * Congenital Diaphragmatic Hernia
  * Heterotaxy
  * Moderate to severe ventriculomegaly or other major brain malformation (not mild isolated ventriculomegaly)
  * Airway obstruction
  * Underlying genetic disease that could impact respiratory function at delivery
  * Arthrogryposis (not apparently isolated clubbed foot)
  * Skeletal dysplasia
* Pregnant patient is unable to understand study materials or is unwilling or unable to consent
* Acute maternal obstetric emergency that precludes time or maternal focus for the consent process to take place

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Number of pre-term neonates that require endotracheal intubation | 30-60 seconds immediately after birth of the newborn
  To determine if deliberate prone positioning of preterm neonates during delayed cord clamping reduces the need for endotracheal intubation in the delivery room.

CONTACTS AND LOCATIONS:
Overall Officials: Katelyn Uribe, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - West Penn Hospital-Allegheny Health Network, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No